CLINICAL TRIAL: NCT01349023
Title: Effects of Energy Density and Energy Content of Pre-portioned entrées on Energy Intake
Brief Title: Energy Content and Energy Density of Pre-portioned Entrees
Acronym: EDEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: FoodED301; R01DK059853 (NIH); R37DK039177 (NIH)
Record Dates: First submitted 2011-05-03; First posted 2011-05-06 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Obesity
Keywords: energy content; energy density; energy intake; pre-portioned entrees
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard Energy content/Standard ED (Experimental)
  Interventions: Other: Energy density (ED), Energy content
- Standard Energy content/Reduced ED (Experimental)
  Interventions: Other: Energy density (ED), Energy content
- Reduced Energy content/Standard ED (Experimental)
  Interventions: Other: Energy density (ED), Energy content
- Reduced Energy content/Reduced ED (Experimental)
  Interventions: Other: Energy density (ED), Energy content

INTERVENTIONS:
Other: Energy density (ED), Energy content — Standard or reduced energy content and energy density of pre-portioned entrees

SUMMARY:
Pre-portioned entrées are commonly consumed to help control portion size and limit energy intake. Few studies, however, have investigated the influence of the characteristics of pre-portioned entrées on energy intake. This study investigates how the characteristics of solid pre-portioned entrées, specifically, variations in their energy content and energy density influence energy intake over a day. The investigators hypothesize that reducing the energy content and energy density of compulsory entrées will act independently and add together to reduce daily energy intake.

DETAILED DESCRIPTION:
This experiment uses a crossover design with repeated measures within subjects. One day a week for four weeks, participants are provided with all of their foods and beverages for breakfast, lunch, and dinner meals. Across test days, the entrée at each meal is varied in both energy content and energy density between a standard level (100%) and a reduced level (64% of the standard). Following consumption of a compulsory entrée, a variety of unmanipulated foods will be served for ad libitum consumption. The order of experimental conditions is counterbalanced across the subjects.

ELIGIBILITY:
Inclusion Criteria:

* regularly eat three meals per day
* do not smoke
* do not have any food allergies or restrictions
* are not athletes in training
* are not dieting
* are not taking medications that would affect appetite
* are willing to consume the foods served in the test meals

Exclusion Criteria:

* a score > 40 on the Zung scale
* a score > 20 on the Eating Attitudes Test
* reported known health problems
* weight not maintained within 10 lb during the 6 months before the start of the study

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Daily Energy Intake (kcal/day) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States